CLINICAL TRIAL: NCT03283215
Title: Causes and Underlying Factors of Faltering Growth Among Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, marina asem shafic, principal investigator, Assiut University
Other Study IDs: IRB00008717
Record Dates: First submitted 2017-08-29; First posted 2017-09-14 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Infants Aged One Month to 2 Years , Infants With Any Type of Feeding (Breast or Artificial or Weaned Attend Assiut University Children Hospital )
MeSH Terms: interventions — Blood Cell Count; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: complete blood count , electrolytes — it is a labarotory test to assess hemoglobin white blood count plate let
  Other Names: urine analysis

SUMMARY:
to research in the different causes of failure to thrive in children including organic and non organic causes

DETAILED DESCRIPTION:
Altered growth velocity in infants has been traditionally described by the term (failure to thrive ) . More recently the preferred terms are faltering growth ,slow weight gain or undernourishment as failure to thrive has been associated with negative connotations of parents failing in their job as careproviders.

The expression 'to falter' means to hesitate. Faltering growth is an observation,without value judgement, of slower than expected rate of growth along an infant's previously defined growth curve.

Faltering growth is a common pediatric problem with many untoward effects . More studies showed that children who failed to thrive in infancy are lighter and shorter at school age with adverse intellectual outcomes (corbett and drewett,2004)(Natale etal., 2014). Weight faltering in the first months of life is particularly associated with these adverse effects.

Infants with faltering growth also have a higher prevalence of feeding problems (Young etal., 2013).Growth failure is more common during infancy than during any other stage of life because programmed growth rates and nutritional needs are high (

ELIGIBILITY:
Inclusion Criteria:

:Infants attending assiut university children hospital who are stunting(decrease height for age ), wasting(decrease weight for lenght ), and underweight (decreases weight for age ) . When all of theses less than -1 Z scores (normal Z-score from -1 to +1 ) . Also mid arm circumference below than 115 mm

Exclusion criteria:

Children complaining of any of the follolowing:

* Malignancy

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants aged 1month upto 2 years infants with any type of feeding (breast , artificial or weaned)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
to recognize nutritional causes of faltering growth | from october 2017 to september 2018
  o recognize nutritional causes of faltering growth by measuring weight ,height ,mid arm circumference ,skin fold thickness